CLINICAL TRIAL: NCT05558228
Title: Accuracy of Doppler Ultrasound Versus Manual Palpation of Pulse in Cardiac Arrest
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Collaborators: Flosonics Medical (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19-0274
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients achieving return of spontaneous circulation: All patients in cardiac arrest with an arterial line in place in the emergency department will be a potential subject. The FloPatch FP120 device will be placed on patients and the carotid artery peak systolic velocity associated with a systolic blood pressure ≥60 mmHg on a femoral arterial line during a pulse check will be determined.
  Interventions: Device: FloPatch FP120
- Patients not achieving return of spontaneous circulation: All patients in cardiac arrest with an arterial line in place in the emergency department will be a potential subject. The FloPatch FP120 device will be placed on patients and the carotid artery peak systolic velocity associated with a systolic blood pressure ≥60 mmHg on a femoral arterial line during a pulse check will be determined.
  Interventions: Device: FloPatch FP120

INTERVENTIONS:
Device: FloPatch FP120 — FloPatch FP120 is an FDA 510(k) cleared device indicated for the non-invasive assessment of blood flow in the carotid artery by medical professionals, such as physicians and nurses. FloPatch uses ultrasound and the Doppler effect to assess blood flow.

SUMMARY:
The FloPatch FP120 device is indicated for use for the noninvasive assessment of blood flow in the carotid artery. The FloPatch FP120 device uses ultrasound and the Doppler effect to non-invasively assess the flow of flood. In this study, the FloPatch FP120 will be applied to the neck at the location of the carotid artery on cardiac arrest patients in the emergency department. FloPatch FP120 data will be compared with arterial line blood pressure to assess for accuracy of pulse checks among cardiac arrest patients in the emergency department.

DETAILED DESCRIPTION:
The FloPatch FP120 device is indicated for use for the noninvasive assessment of blood flow in the carotid artery. The FloPatch FP120 device uses ultrasound and the Doppler effect to non-invasively assess the flow of flood. In this study, the FloPatch FP120 will be applied to the neck at the location of the carotid artery on cardiac arrest patients in the emergency department. This study will determine the peak systolic velocity, as measured by the FLoPatch FP120 device, that is associated with a systolic blood pressure of ≥60 mmHg on a femoral arterial line in cardiac arrest patients during a pulse check. The associated accuracy, sensitivity, and specificity of the calculated pulse systolic velocity to detect return of spontaneous circulation with a systolic blood pressure ≥60 mmHg in cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* In cardiac arrest at the North Shore University Hospital emergency department
* Arterial line placed during cardiac arrest resuscitation

Exclusion Criteria:

* Traumatic cardiac arrest
* Patients without bilateral lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18+ years of age in atraumatic cardiac arrest with an arterial line placed in the emergency department during resuscitation.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-09-06 (Estimated); Study Completion 2024-09-06 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Return of Spontaneous Circulation | 30 minutes
  Any patient achieving any episode of return of spontaneous circulation during a pulse check will be considered as having the outcome. Cardiac arrest resuscitations are typically not longer than 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Cohen, MD, Principal Investigator — North Shore University Hospital
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No